CLINICAL TRIAL: NCT03312556
Title: Treatment of Supine Hypertension in Autonomic Failure With Continuous Positive Airway Pressure
Brief Title: Treatment of Supine Hypertension in Autonomic Failure (CPAP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 010189-1; 200124 (Other: Vanderbilt IRB)
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Supine Hypertension; Autonomic Failure
Keywords: hypertension; supine hypertension; autonomic failure; pure autonomic failure; multiple system atrophy; cpap
MeSH Terms: conditions — Pure Autonomic Failure; Hypertension; Multiple System Atrophy; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Placebo pill or patch or sham CPAP (Placebo Comparator): Placebo pill or patch or sham CPAP
  Interventions: Drug: Placebo
- CPAP (continuous positive airway pressure) (Active Comparator): Continuous positive airway pressure during the night
  Interventions: Device: continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: continuous positive airway pressure (CPAP) — Continuous positive airway pressure(CPAP) will be applied during the night starting from 20:00. CPAP level will be determined during an acute CPAP trial.
  Other Names: CPAP
  Arms: CPAP (continuous positive airway pressure)
Drug: Placebo — Placebo pill or patch. Single dose
  Other Names: placebo pill or patch
  Arms: Placebo pill or patch or sham CPAP

SUMMARY:
Supine hypertension is a common problem that affects at least 50% of patients with primary autonomic failure. Supine hypertension can be severe and complicates the treatment of orthostatic hypotension. The purpose of this study is to assess whether continuous positive airway pressure (CPAP) decreases blood pressure in autonomic failure patients with supine hypertension.

DETAILED DESCRIPTION:
Supine hypertension is a common problem that affects at least 50% of patients with primary autonomic failure. Supine hypertension can be severe and complicates the treatment of orthostatic hypotension. Drugs used for the treatment of orthostatic hypotension (eg, fludrocortisone and pressor agents), worsen supine hypertension. High blood pressure may also cause target organ damage in this group of patients. The pathophysiologic mechanisms causing supine hypertension in patients with autonomic failure have not been defined.

This study will test the hypothesis that continuous positive airway pressure (CPAP) has an acute lowering-BP effect in autonomic failure patients with supine hypertension. CPAP is a widely-used treatment for sleep-related breathing disorders including sleep apnea, that uses mild air pressure to keep the breathing airways open. It involves using a CPAP machine that blows air into a tube connected to a mask placed over the nose, or nose and mouth. For these studies, a commercial CPAP device will be used to apply pressure sequentially at 0, 4, 8, 12 and 16 cm H2O for 1-20 minute each. Depending on the BP response and tolerability to CPAP, CPAP may be applied during the night using a CPAP level that was tolerable and showed a BP-lowering effect during the acute test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with autonomic failure and with supine hypertension from all races

Exclusion Criteria:

* All medical students
* Pregnant women
* High-risk patients (e.g. heart failure, symptomatic coronary artery disease, liver impairment, history of stroke or myocardial infarction)
* History of serious allergies or asthma.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-12-21 (Estimated)

PRIMARY OUTCOMES:
Supine Systolic Blood Pressure | 12 hours
  change in supine systolic blood pressure from baseline

SECONDARY OUTCOMES:
Urinary volume | 12 hours
  Nocturnal urinary volume

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center/ Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okamoto LE, Celedonio JE, Smith EC, Paranjape SY, Black BK, Wahba A, Park JW, Shibao CA, Diedrich A, Biaggioni I. Continuous Positive Airway Pressure for the Treatment of Supine Hypertension and Orthostatic Hypotension in Autonomic Failure. Hypertension. 2023 Mar;80(3):650-658. doi: 10.1161/HYPERTENSIONAHA.122.20081. Epub 2023 Jan 5. PMID 36601916